CLINICAL TRIAL: NCT05172037
Title: An Adaptive, Multicenter, Randomized, Double-blind, Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of Aerosolized JH509 vs. Placebo in Non-hospitalized Adult Patients With Mild COVID-19
Brief Title: Novaferon in Non-hospitalized Adult Patients With Mild COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genova Inc. (Industry)
Collaborators: Tokyo Shinagawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JH-COR-007
Record Dates: First submitted 2021-12-26; First posted 2021-12-29 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Covid19
Keywords: antiviral; SARS-CoV-2; COVID19
MeSH Terms: conditions — COVID-19 | interventions — recombinant interferon alpha 2b-like protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novaferon (Active Comparator): Inhaled Novaferon, given 20 ug BID, daily for 7 days
  Interventions: Biological: Novaferon
- Placebo (Placebo Comparator): Inhaled saline (placebo), given BID, daily for 7 days
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Novaferon — a novel recombinant antiviral protein drug
  Arms: Novaferon
Biological: Placebo — Saline
  Arms: Placebo

SUMMARY:
An Adaptive, Multicenter, Randomized, Double-blind, Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of Aerosolized JH509 vs. Placebo in Non-hospitalized Adult Patients with Mild COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from the participants with an age of over 20 years at the time of signing the informed consent.
2. SARS-CoV-2 infection is diagnosed by RT-PCR within 72 hours before starting drug administration.
3. Less than six days from onset of COVID-19-related symptoms below to starting the administration of the investigational drug with at least one of the following symptoms observed at the time of enrollment : fever (37.5C or higher), respiratory symptoms (cough, shortness of breath, sore throat, runny nose, etc.), headache, myalgia, malaise, abdominal pain, diarrhea, nausea/vomiting, dysosmia, dysgeusia, or other COVID-19 symptoms defined by investigators or coinvestigators investigators.
4. Oxygen saturation (SpO2) measured by pulse oximeter is more than 95%.
5. Require no supplemental oxygen.
6. Women (less than 12 months after the last menstrual period) who have a negative pregnancy test (urine hCG qualification) and agree to use highly effective contraceptive methods (taking oral contraceptives or use of condom by male partner) during the study period. Investigators or coinvestigators investigators will provide guidance on contraceptive methods.
7. Women who are not breast-feeding.

Exclusion Criteria:

1. History of hypersensitivity to interferon or JH509 or any excipients of interferon or JH509.
2. Have received antiviral treatments and drugs expected to have antiviral effects (Favipiravir, Remdesivir, Interferon, Nafamostat mesilate, and Basiliximab/Imdevimab, including drugs that are being newly developed and that have been approved) in the past or having had it considered necessary to receive these treatments during the study period.
3. Having had it considered necessary to receive treatments, such as drugs containing corticosteroids (excluding topical drugs), antimicrobial agents, and inhalants other than the investigational drug during the study period.
4. Taking "Shosaikoto," an herbal medicine.
5. Neuropsychiatric disorder and autoimmune disorder.
6. CTCAE Grade 3 or higher liver dysfunction (ALT/AST > 5ULN) or renal dysfunction (eGFR < 30 mL/min/1.73 m2).
7. Active infections or other medical conditions that contraindicate inhalation therapy.
8. Having the complication of malignant tumor or a history of malignant tumor within 1 year before consent acquisition.
9. Inappropriate for inclusion in the clinical trial as determined by investigators or coinvestigators investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 222 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Rate of severe conditions with Score 3 or more serious on a seven-point ordinal scale from the start date of investigational drug administration (Day 1) to Day 28. | 28 day

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo Shinagawa Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No